CLINICAL TRIAL: NCT00927836
Title: AXIS 2: AX200 for the Treatment of Ischemic Stroke - A Multinational, Multicenter, Randomized, Doubleblind, Placebo-controlled Phase II Trial
Brief Title: AXIS 2: AX200 for the Treatment of Ischemic Stroke
Acronym: AXIS-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sygnis Bioscience GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AX200-101; EudraCT 2008-006444-19
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-08

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Filgrastim; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AX200 (Experimental)
  Interventions: Biological: Filgrastim
- Placebo (Placebo Comparator)
  Interventions: Drug: Sodium chloride solution

INTERVENTIONS:
Biological: Filgrastim — 135 μg/kg body weight total dose Short term infusion (20 to 30 minutes) and continuous infusion over 3 days
  Arms: AX200
Drug: Sodium chloride solution — Short term infusion (20 to 30 minutes) and continuous infusion over 3 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of AX200 (filgrastim) in the treatment of acute ischemic stroke and to assess the safety and tolerability of AX200.

ELIGIBILITY:
Major Inclusion Criteria:

* diagnosis of acute ischemic stroke with an onset within 9 hours prior to start of study agent administration
* ischemic stroke in the MCA territory confirmed by MRI (diffusion)
* age ≥18 years and ≤85 years
* lesion size on DWI ≥15 ccm
* written informed consent

Major Exclusion Criteria:

* prior to current stroke: inability to walk or to lead an independent life
* life expectancy less or equal 6 months
* stupor or coma
* lacunar infarct
* any evidence of ICH
* malignant hypertension
* presence of history of active malignancies
* platelet count <100/nl at randomization
* leukocyte count >20/nl at randomization
* congenital neutropenia
* pregnant or lactating women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2009-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Improvement on mRS relative to placebo-treated patients | day 90

SECONDARY OUTCOMES:
Improvement on NIHSS relative to placebo-treated patients | day 90

CONTACTS AND LOCATIONS:
Overall Officials: Frank Rathgeb, Dr., Study Chair — Sygnis Bioscience GmbH & Co KG; Rico Laage, Dr., Study Director — Sygnis Bioscience GmbH & Co KG
Locations (58):
- Austria (3):
  - Landes-Nervenklinik Wagner-Jauregg, Linz
  - AHK Linz, Linz
  - Wilhelminenspital, Vienna
- Belgium (4):
  - AZ Sint-Jan AV, Bruges
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Gasthuisberg, Leuven
- Czechia (7):
  - St. Anne's Faculty Hospital, Brno
  - Faculty Hospital, Olomouc
  - Faculty Hospital Ostrava, Ostrava
  - Municipal Hospital Ostrava, Ostrava
  - Faculty Hospital 1, Plzeň - Lochotín
  - General Faculty Hospital, Prague
  - Faculty Hospital Motol, Prague
- Germany (24):
  - Universitätsklinikum der RWTH Aachen, Aachen
  - Kreiskrankenhaus Altenburg gGmbH, Altenburg
  - Charité Universitätsmedizin Berlin, Berlin
  - Charite Universitätsklinikum "Benjamin Franklin" Klinik und Poliklinik für Neurologie, Berlin
  - Evangelisches Krankenhaus Bielefeld, Bielefeld
  - Klinikum Bremen-Mitte gGmbH, Bremen
  - Klinik für Neurologie Chemnitz, Chemnitz
  - Marienhospital Düsseldorf, Düsseldorf
  - Universität Erlangen-Nürnberg, Erlangen
  - Universitätsklinikum Essen, Essen
  - Neurologische Universitätsklinik Freiburg, Freiburg im Breisgau
  - Berufsgenossenschaftliche Kliniken Bergmannstrost, Halle
  - Universitätsklinik Hamburg Eppendorf, Hamburg
  - Universität Heidelberg, Heidelberg
  - Friedrich-Schiller-Universitätsklinikum, Jena
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum der Stadt Ludwigshafen, Ludwigshafen
  - Philipps-Universität Marburg, Marburg
  - Technische Universität München Klinikum rechts der Isar, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Osnabrück GmbH, Osnabrück
  - Asklepios Fachklinikum Teupitz, Teupitz
  - Neurologische Klinik, Eberhard-Karls-Universität Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Poland (5):
  - Klinika Neurologii z Pododdziałem Udarowym, Bialystok
  - Wojewódzki Szpital Specjalistyczny im. Mikołaja Kopernika w Gdańsku, Oddział Neurologiczny i Leczenia Udarów Mózgu, Gdansk
  - Uniwersytecki Szpital Kliniczny im. Wojskowej Akademii Medycznej Uniwersytetu Medycznego w Łodzi, Centralny Szpital Weteranów, Klinika neurologii i epileptologii z oddziałem udarowym, Lodz
  - II Klinika Neurologii, Warsaw
  - Instytut Psychiatrii i Neurologii, I Klinika neurologii, Warsaw
- Slovakia (7):
  - Comenius University Bratislava, Bratislava
  - 4. Faculty Hospital with Policlinic, Bratislava
  - Faculty Hospital L. Derer, Bratislava
  - Faculty Hospital, Košice
  - Faculty Hospital, Martin
  - Faculty Hospital Nitra, Nitra
  - Fakultna nemocnica Trnava, Trnava
- Spain (8):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Dr. Josep Trueta, Girona
  - Hospital de la Princesa, Madrid
  - Hospital Ramon y Cajal / Fundacion para le Investigacion Biomedica del Hospital Ramon y Cajal, Madrid
  - Hopsital Univ. La Paz / Fundacion para la Investigacion, Madrid
  - Hospital Univ. Virgen del Rocio, Seville
  - Hospital Clínico Universitario, Valencia

REFERENCES:
- [Derived] Scheldeman L, Wouters A, Dupont P, Christensen S, Boutitie F, Cheng B, Ebinger M, Endres M, Fiebach JB, Gerloff C, Muir KW, Nighoghossian N, Pedraza S, Simonsen CZ, Ringelstein EB, Chamorro A, Grond M, Laage R, Schneider A, Thomalla G, Thijs V, Lemmens R. Reversible Edema in the Penumbra Correlates With Severity of Hypoperfusion. Stroke. 2021 Jul;52(7):2338-2346. doi: 10.1161/STROKEAHA.120.033071. Epub 2021 May 13. PMID 33980046
- [Derived] Bu N, Khlif MS, Lemmens R, Wouters A, Fiebach JB, Chamorro A, Ringelstein EB, Norrving B, Laage R, Grond M, Wilms G, Brodtmann A, Thijs V. Imaging Markers of Brain Frailty and Outcome in Patients With Acute Ischemic Stroke. Stroke. 2021 Mar;52(3):1004-1011. doi: 10.1161/STROKEAHA.120.029841. Epub 2021 Jan 28. PMID 33504185
- [Derived] Kufner A, Wouters A, Bracoud L, Laage R, Schneider A, Schabitz WR, Hermier M, Thijs V, Fiebach JB; AXIS2 investigators. Infarct volume-based subgroup selection in acute ischemic stroke trials. Stroke. 2015 May;46(5):1368-70. doi: 10.1161/STROKEAHA.114.008115. Epub 2015 Mar 12. PMID 25765724
- [Derived] Ringelstein EB, Thijs V, Norrving B, Chamorro A, Aichner F, Grond M, Saver J, Laage R, Schneider A, Rathgeb F, Vogt G, Charisse G, Fiebach JB, Schwab S, Schabitz WR, Kollmar R, Fisher M, Brozman M, Skoloudik D, Gruber F, Serena Leal J, Veltkamp R, Kohrmann M, Berrouschot J; AXIS 2 Investigators. Granulocyte colony-stimulating factor in patients with acute ischemic stroke: results of the AX200 for Ischemic Stroke trial. Stroke. 2013 Oct;44(10):2681-7. doi: 10.1161/STROKEAHA.113.001531. Epub 2013 Aug 20. PMID 23963331